CLINICAL TRIAL: NCT01596452
Title: Enumeration of Circulating Tumour Cells (CTCs) in Patients With Advanced Solid Malignancy Using Complementary Metal Oxide Semiconductor (CMOS) Technology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: Version 1
Record Dates: First submitted 2012-04-02; First posted 2012-05-11 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Modern anti-cancer treatments are focused on development of molecular based therapies i.e. specific treatments targeted against underlying biological processes. There is still much to learn about the biology of cancer, especially in tumours such as colorectal and lung cancer where it is likely multiple heterogenous signaling pathways are responsible for progression of disease. This project aims to evaluate circulating tumour cells (CTCs) as a surrogate biomarker for tumour characteristics and to determine how they may used to identify new targets for therapeutic agents. Their use could be applied to diagnosis of cancer, prediction of response to therapies and prognosis, ultimately across a broad range of tumour types. Currently the only way to investigate molecular features of a cancer is through procurement of an invasive tumour biopsy that is often difficult to obtain, often results in insufficient material and is unpleasant for the patient. A blood-based test would provide a much more practical and patient friendly alternative. The enumeration and molecular characterisation of CTCs has the novel potential of being a "virtual biopsy" of the tumour and offers the opportunity for immediate therapeutic decisions (eg. if the tumour develops a therapy resistant genotype while on treatment). CTCs have been known to circulate in bloodstream of cancer patients for many years and are known to lead to cancer metastases. They have been very difficult to detect, up until recently, due to the complexity of the metastatic process and detecting relatively small numbers of CTCs amongst billions of red and white blood cells. However, technology has moved on dramatically in the last few years. The FDA approved CellSearch platform (Veridex, NJ) can isolate and enumerate CTCs based on the immunomagnetic capture of EpCAM (epithelial cell adhesion molecule) positive cells. Several studies have recently demonstrated the value of CTC enumeration in reflecting prognosis and predicting early response to systemic chemotherapy. For example, in a study comprising 456 patients with metastatic colorectal cancer starting a new line of therapy, patients with =3 CTCs per 7.5 ml blood at baseline had shorter progression free survival (PFS) and overall survival (OS) compared to those patients with < 3CTCs at baseline (PFS 4.5 versus 7.9 months P=0.0001; OS 8.5 versus 19.1 months P=0.0000 respectively). Overall survival for patients converting to or maintaining CTCs =3 within a few weeks of commencing systemic therapy remained worse than for those patients maintaining CTC counts < 3 per 7.5ml blood. Similar results have been reported in patients with breast and hormone refractory prostate cancer (HRPC). These studies have led to FDA approval of the CellSearch system as an adjunct to monitoring patients with these 3 tumour types. The CellSearch platform, however, does not allow for the downstream DNA analysis of captured cells and the ferroparticle-coated CTCs are non-viable. Furthermore, this platform is a multi-machine, multi-kit system that is laborious (typical 3-7 days turnover time), expensive (USD 650), and subject to operator variance. In this protocol, the investigators propose for the first time, an automated, fully quantitative system for isolation and enrichment of CTCs. The key differentiating feature of our novel CMOS system is the electrochemical identification and counting of tumour cells using a high density electrode array with associated electronics for addressing the electrodes. This leads to a standardized assay for tumour cells with a shorter turnover time and without the need of a skilled operator. This system also holds the potential for allowing the molecular characterization of CTCs. This study aims to enumerate CTCs using a novel CMOS technology in patients with metastatic cancer who are scheduled to receive palliative chemotherapy, and to correlate CTC number with clinical outcome. In Part I of the study, the investigators will recruit 10 patients with metastatic NSCLC and 10 patients with metastatic CRC in order to assess the feasibility of CTC enumeration in patients. In particular, the investigators aim to establish whether CTCs are detectable using the novel CMOS technology in patients with metastatic cancer. In Part II of the study, the investigators will recruit 21 patients with metastatic NSCLC and 89 patients with metastatic CRC in order to compare CTC counts as determined by the CMOS technology with CTC counts as determined by the CellSearch platform. Blood samples will be collected at a single time point prior to the start of palliative chemotherapy. CTC numbers will be correlated with clinical outcome in all evaluable patients.

The investigators hypothesize that CTC enumeration by a novel CMOS technology is non-inferior to CTC enumeration by the CellSearch platform in patients with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of either metastatic NSCLC or metastatic CRC are eligible.
2. Patients should be due to undergo palliative chemotherapy as part of their standard clinical care.
3. Patients must be able to receive and understand verbal and written information regarding the study and give written, informed consent.

Exclusion Criteria:

1. Persons under 18 years of age.
2. Conditions in which research blood sampling may increase risk of complications for the patient and/or the investigators. For example, uncontrolled bleeding, patients with a known blood-borne viral infection (eg. hepatitis B or C, HIV) or poor venous access.
3. Other persons in whom clinical judgement by the investigator concluded that the patient should not participate in the study. For example, anticipated poor compliance to attend for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated for cancer at the National University Hospital (NUH), Singapore
Sampling Method: Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Establish whether CTCs are detectable using novel CMOS technology in patients with metastatic cancer. | 1 year

SECONDARY OUTCOMES:
Compare CTC counts as determined by CMOS technology with CTC counts as determined by immunomagnetic capture with the CellSearch platform (Veridex, NJ). | 1 year
Determine the relationship between baseline CTC number as determined by CMOS technology and clinical outcome. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ying Kiat Zee, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Cristofanilli M, Budd GT, Ellis MJ, Stopeck A, Matera J, Miller MC, Reuben JM, Doyle GV, Allard WJ, Terstappen LW, Hayes DF. Circulating tumor cells, disease progression, and survival in metastatic breast cancer. N Engl J Med. 2004 Aug 19;351(8):781-91. doi: 10.1056/NEJMoa040766. PMID 15317891
- [Background] Cristofanilli M, Hayes DF, Budd GT, Ellis MJ, Stopeck A, Reuben JM, Doyle GV, Matera J, Allard WJ, Miller MC, Fritsche HA, Hortobagyi GN, Terstappen LW. Circulating tumor cells: a novel prognostic factor for newly diagnosed metastatic breast cancer. J Clin Oncol. 2005 Mar 1;23(7):1420-30. doi: 10.1200/JCO.2005.08.140. PMID 15735118